CLINICAL TRIAL: NCT04107246
Title: Data Collection of Therapeutic Compliance in Patients Receiving Corneal Graft Using a Collection Box for Corticosteroid Eye Drops
Acronym: KALICORT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Kali Care (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19CH145; 2019-A02280-57 (Other: ANSM)
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Corneal Graft Disorder (Disorder); Corticosteroid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly transplanted corneal patients
  Interventions: Device: use of the KaliJAR box

INTERVENTIONS:
Device: use of the KaliJAR box — KaliJAR® : validated device for single-dose eye drops collection. the patient will be asked to discard each single dose of eye drops in the KaliJAR box. The patient returns with the KaliJAR box at each consultation as part of normal practice. The KaliJAR box will be emptied at each consultation by the doctor and then returned to the patient.
  No further examination or visit.

SUMMARY:
Following corneal graft, local steroids with a gradually decreasing dose for 12 months are prescribed to reduce the graft rejection risk (maximum incidence of 20% for the first 12 months). The validated KaliJAR® device is a box for single-dose eye drops collection. This innovative tool will make it possible to objectify the compliance of patients with a corneal graft.

Unlike the field of glaucoma, no specific compliance data are available for corneal grafts, although it is important because graft rejection is the most important cause of corneal graft failure.

ELIGIBILITY:
Inclusion Criteria:

* Newly transplanted corneal patients
* Patients able to instill correctly topical corticosteroid treatment
* Patients able to come to control visits
* Patient affiliated or entitled to a social security system
* Patient informed about the study and having signed a consent

Exclusion Criteria:

* Patients under guardianship
* Patients unable to give their consent or to correctly use the collection box

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly transplanted corneal patients and adult
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Ratio between the number of instilled drops / number of prescribed drops | 12 months

SECONDARY OUTCOMES:
patient behaviour towards corticosteroid treatment | 12 months
  Compliance curve for each patient (pattern / compliance pattern). Compliance profiles versus prescribed treatment at fixed interval time
Questionnaire on therapeutic compliance | month 1, month 6 and month 12
  Morisky questionnaire :
  Adherence to treatment is good if the score is greater than or equal to 8. Adherence to treatment is average if the score is 6 or 7. Adherence to treatment is low if the score is less than 6.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GAIN, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No